CLINICAL TRIAL: NCT02206425
Title: A Phase 1/2 Study of Ixazomib as a Replacement for Bortezomib or Carfilzomib for Multiple Myeloma (MM) Patients Recently Relapsed or Refractory to Their Last Combination Regimen Containing Either Bortezomib or Carfilzomib
Brief Title: Ixazomib as a Replacement for Carfilzomib and Bortezomib for Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X16041; IISR-2013-M100118 (Other: Takeda)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Relapsed/refractory; Ixazomib; Proteasome inhibitor; Oral
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Melphalan; Prednisone; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Ascorbic Acid; 1-dodecylpyridoxal; liposomal doxorubicin; Doxorubicin; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- bortezomib + melphalan + prednisone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Melphalan; Drug: Prednisone
- bortezomib + dexamethasone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone
- carfilzomib + dexamethasone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone
- bortezomib + lenalidomide + dexamethasone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide
- carfilzomib + lenalidomide + dexamethasone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide
- bortezomib + cyclophosphamide + dexamethasone (Experimental): MTD determination. Ixazomib will be administered on Days 1, 8 and 15 of a 28-day cycle at a starting dose of 3 mg in Cycle 1, and then intra-patient dose-escalation will proceed to 4 mg in Cycle 2. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone
- bortezomib + cyclophosphamide + ascorbic acid (Experimental): MTD determination. Ixazomib will be administered on Days 1, 8 and 15 of a 28-day cycle at a starting dose of 3 mg in Cycle 1, and then intra-patient dose-escalation will proceed to 4 mg in Cycle 2. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib. Due to a potential drug-drug interaction between ixazomib and ascorbic acid, patients will receive ixazomib in the clinic in the morning and will be instructed to take ascorbic acid in the evening, followed by cyclophosphamide.
  Interventions: Drug: Cyclophosphamide; Dietary Supplement: Ascorbic acid
- bortezomib + PLD + dexamethasone (Experimental): MTD determination. Ixazomib will be administered on Days 1, 8 and 15 of a 28-day cycle at a starting dose of 3 mg in Cycle 1, and then intra-patient dose-escalation will proceed to 4 mg in Cycle 2. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone; Drug: PLD
- bortezomib + pomalidomide + dexamethasone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone; Drug: Pomalidomide
- carfilzomib + pomalidomide + dexamethasone (Experimental): Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed. Patients that were on a 21-day cycle schedule will follow a 28-day cycle schedule and receive ixazomib on days 1, 8 and 15. Other drugs will be administered on the same days as they were given on their prior 21-day cycle schedule, except that, in the new 28-day schedule, day 1 of other drugs will be the same as day 1 of ixazomib.
  Interventions: Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Melphalan — Melphalan will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Phenylalanine mustard; Alkeran
  Arms: bortezomib + melphalan + prednisone
Drug: Prednisone — Prednisone will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Cortan; Deltasone; Orasone; Prednisone Intensol; Sterapred; Sterapred DS
  Arms: bortezomib + melphalan + prednisone
Drug: Cyclophosphamide — Cyclophosphamide will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Cytoxan; CPM; CTX; CYT
  Arms: bortezomib + cyclophosphamide + ascorbic acid; bortezomib + cyclophosphamide + dexamethasone
Drug: Dexamethasone — Dexamethasone will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Decadron; Dexamethasone Intensol; Dexpak Taperpak
  Arms: bortezomib + PLD + dexamethasone; bortezomib + cyclophosphamide + dexamethasone; bortezomib + dexamethasone; bortezomib + lenalidomide + dexamethasone; bortezomib + pomalidomide + dexamethasone; carfilzomib + dexamethasone; carfilzomib + lenalidomide + dexamethasone; carfilzomib + pomalidomide + dexamethasone
Dietary Supplement: Ascorbic acid — Vitamin C will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Vitamin C
  Arms: bortezomib + cyclophosphamide + ascorbic acid
Drug: PLD — Pegylated liposomal doxorubicin will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: ATI-0918; doxorubicin hydrochloride liposome; doxorubicin hydrochloride liposome injection; liposomal adriamycin; liposomal doxorubicin; liposomal doxorubicin hydrochloride; liposome-encapsulated doxorubicin; pegylated doxorubicin HCl liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; DOXIL; Dox-SL; Evacet; LipoDox
  Arms: bortezomib + PLD + dexamethasone
Drug: Lenalidomide — Lenalidomide will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Revlimid
  Arms: bortezomib + lenalidomide + dexamethasone; carfilzomib + lenalidomide + dexamethasone
Drug: Pomalidomide — Pomalidomide will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed (it varies with each patient).
  Other Names: Pomalyst
  Arms: bortezomib + pomalidomide + dexamethasone; carfilzomib + pomalidomide + dexamethasone

SUMMARY:
The goal of this clinical research study is to evaluate the safety and effectiveness (good and bad effects) of ixazomib given as part of a combination therapy to treat subjects with relapsed (subjects whose disease came back) or refractory (subjects whose disease did not respond to past treatment) multiple myeloma. More specifically, the study is focused on subjects who were previously treated with bortezomib (Velcade®) or carfilzomib (Kyprolis®) and showed worsening of their myeloma while receiving either one of these drugs in combination therapy. This study is a Phase I/II. Ixazomib is an investigational drug, which means that ixazomib is currently being tested and is not yet approved by the United States Food and Drug Administration (FDA) for subjects with relapsed or refractory multiple myeloma. Ixazomib is a new study drug that belongs to the same class as bortezomib and carfilzomib; however, unlike bortezomib and carfilzomib, ixazomib is taken by mouth. Current studies investigating ixazomib are demonstrating that it is as safe as bortezomib and effective for the treatment of multiple myeloma both on its own and in combination with other multiple myeloma medications, such as lenalidomide and dexamethasone, or prednisone and melphalan.

DETAILED DESCRIPTION:
This is a phase 1/2, intra-patient, multicenter, open-label and non-randomized study to evaluate the efficacy and safety of ixazomib as a replacement for bortezomib or carfilzomib among multiple myeloma (MM) patients who have failed proteasome inhibitor (PI)-containing combination regimens. Patients will receive ixazomib once a week in place of bortezomib or carfilzomib in combination with an alkylating agent (melphalan or cyclophosphamide), anthracycline (pegylated doxorubicin [PLD]), immunomodulatory agent (lenalidomide, pomalidomide), ascorbic acid and/or a glucocorticosteroid (dexamethasone, prednisone or methylprednisolone) administered using the same dose(s) and schedule(s) as the last PI-containing regimen that the patients had received and failed. The total number of different prior bortezomib- or carfilzomib-containing regimens that will be evaluated is 10, reflecting those commonly used in the community as follows:

* bortezomib + melphalan + prednisone
* bortezomib + cyclophosphamide + ascorbic acid
* bortezomib + cyclophosphamide + dexamethasone
* bortezomib + PLD + dexamethasone
* bortezomib + dexamethasone
* carfilzomib + dexamethasone
* bortezomib + lenalidomide + dexamethasone
* bortezomib + pomalidomide + dexamethasone
* carfilzomib + lenalidomide + dexamethasone
* carfilzomib + pomalidomide + dexamethasone

This study will enroll 60 patients who are refractory to a bortezomib- or carfilzomib-containing combination regimen, as demonstrated by progressive disease (PD) while being treated, or who have relapsed within 8 weeks from the last dose of bortezomib or carfilzomib in their last PI-containing combination regimen.

Ixazomib will replace bortezomib or carfilzomib using the same PI-containing regimen the patients failed.The study will consist of: 1) a screening period; 2) up to eight 28-day treatment cycles; 3) a maintenance period; 4) a final assessment to occur 28 days after the end of the last treatment cycle; and 5) a follow-up period.

Ixazomib will be administered PO at 4 mg on Days 1, 8 and 15 of a 28-day cycle to patients enrolled in seven regimens (bortezomib + melphalan + prednisone, bortezomib + dexamethasone, carfilzomib + dexamethasone, bortezomib + lenalidomide + dexamethasone, bortezomib + pomalidomide + dexamethasone, carfilzomib + lenalidomide + dexamethasone, carfilzomib + pomalidomide + dexamethasone). Subjects on those regimens receiving 4 mg of ixazomib from the beginning of the trial will continue to do so for the length of the study, unless they suffer from adverse events requiring dose reductions. For the other three regimens, bortezomib + cyclophosphamide + dexamethasone, bortezomib + cyclophosphamide + ascorbic acid, and bortezomib + PLD + dexamethasone, the MTD for ixazomib is unknown and intra-patient dose escalation will be performed to determine the specific MTD for each of them. For these three regimens, ixazomib will be administered on Days 1, 8 and 15 of a 28-day cycle at a starting dose of 3 mg in Cycle 1, and then intra-patient dose-escalation will proceed to 4 mg in Cycle 2. All other agents will be administered at the same schedule and dose intensity as those of the last PI-containing treatment the patient failed.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients 18 years or older
2. Patients must have a diagnosis of MM, based on standard criteria as follows:

   * Major criteria:

     1. plasmacytomas on tissue biopsy
     2. bone marrow plasmacytosis (greater than 30% plasma cells)
     3. monoclonal immunoglobulin spike on serum electrophoresis IgG greater than 3.5 g/dL or IgA greater than 2.0 g/dL; kappa or lambda light chain excretion greater than 1 g/day on 24 hour urine protein electrophoresis
   * Minor criteria:

     1. bone marrow plasmacytosis (10% to 30% plasma cells)
     2. monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
     3. lytic bone lesions
     4. normal IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL

   Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:
   * any 2 of the major criteria
   * major criterion 1 plus minor criterion 2, 3, or 4
   * major criterion 3 plus minor criterion 1 or 3
   * minor criteria 1, 2, and 3, or 1, 2, and 4
3. Currently has progressive MM that has previously progressed or is currently progressing while receiving or within 8 weeks of receiving bortezomib or carfilzomib as part of a combination treatment. MM patients that demonstrate refractory disease, as defined below, are both eligible for enrollment provided they fulfill the other eligibility criteria:

   • Patients are refractory to a bortezomib or carfilzomib combination regimen, when they progress while currently receiving a bortezomib or carfilzomib combination treatment, or within 8 weeks of its last dose. Patients are considered relapsed, when they progress between 8 and 12-weeks from their last dose of bortezomib or carfilzomib as part of a bortezomib or carfilzomib combination therapy. Prior treatment with four days or less of a total of 400 mg of prednisone (or an equivalent potency of another steroid) for MM will not be considered a regimen.
4. Patients that were on bortezomib-containing regimens must have been administered at least 4 doses of a minimum of 1.0 mg/m2 in no more than 28-days cycles. Subjects must have received at least one cycle meeting this definition and have shown PD to be considered eligible
5. Patients that were on carfilzomib-containing regimens must have received at least 6 doses of at least 27 mg/m2 in no more than 28 days per cycle. Subjects must have received at least one cycle meeting this definition and have shown PD to be considered eligible
6. Progressed from one of the specific bortezomib- or carfilzomib-containing regimens as listed on page 51. Although bortezomib- and carfilzomib-containing combination regimens that are otherwise identical except for the PI result in the same ixazomib regimen, they will be enrolled separately so that safety/efficacy can be separately determined, thereby allowing comparisons based on the prior PI that subjects were exposed to as part of the regimen that they failed (carfilzomib vs. bortezomib)
7. Patient may have received a carfilzomib- or bortezomib-containing regimen at any time and may have received other non-proteasome inhibitor-containing intervening treatments

Key Exclusion Criteria:

1. Patient has been diagnosed with:

   1. Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M protein) and skin changes (POEMS) syndrome.3
   2. Primary amyloidosis
   3. Plasma cell leukemia
   4. Severe hypercalcemia, i.e., serum calcium = 12 mg/dL (3.0 mmol/L) corrected for albumin
2. Diagnosed or treated for another malignancy within 3 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanomatous skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. Impaired cardiac function or clinically significant cardiac diseases, including myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, clinically significant pericardial disease, severe uncontrolled ventricular arrhythmias, echocardiogram or multigated acquisition scan (MUGA) evidence of left ventricular ejection fraction (LVEF) below institutional normal within 28 days prior to enrollment, electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant
4. Patient has peripheral neuropathy grade 3 or higher or Grade 2 with pain on clinical examination during the screening period
5. Patient has received the following prior therapy:

   1. Chemotherapy within 21 days of enrollment (6 weeks for nitrosoureas)
   2. Corticosteroids (>10 mg/day prednisone or equivalent) within 21 days of enrollment
   3. Immunotherapy or antibody therapy as well as thalidomide, pomalidomide, lenalidomide, arsenic trioxide, carfilzomib, or bortezomib within 21 days before enrollment
6. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
7. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for selected regimens | Cycles 1-2 for selected regimens (up to 2 months)
  MTD determined via the number of dose-limiting toxicities (DLTs) per cohort for the following ixazomib- containing combinations:
  bortezomib+ cyclophosphamide + dexamethasone, bortezomib + cyclophosphamide + ascorbic acid, bortezomib + PLD + dexamethasone
Number of subjects with adverse events | up to 48 months
  Occurrence of adverse events throughout the study, graded via CTCAE v 4.03 criteria
Overall response rate (ORR) | up to 48 months
  Complete response (CR)+ very good partial response (VGPR) + partial response (PR), defined using IMWG criteria
Clinical benefit rate (CBR) | up to 48 months
  CBR=ORR + minor response (MR)

SECONDARY OUTCOMES:
Time to Progression | at least over 48 months
  Time from initiation of therapy to progressive disease
Progression-free survival (PFS) | at least over 48 months
  Time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
Time to response (TTR) | up to 48 months
  Time from the initiation of therapy to the first evidence of a confirmed response
Duration of response (DOR) | at least over 48 months
  Time from the first response (> PR) to progressive disease
Overall survival (OS) | at least over 48 months
  Time from initiation of therapy to death from any cause or last follow-up visit
Peripheral Neuropathy (PN) | up to 48 months
  Incidence and severity among patients receiving ixazomib compared to their baseline PN when they entered the trial, defined by CTCAE v4.0.3 and FACT-GOG/NTX questionnaire score.

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — James R. Berenson MD, Inc.
Locations (12):
- United States (12):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - John Muir Health Clinical Research Center, Concord, California
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - Robert A. Moss, MD, FACP, Inc, Fountain Valley, California
  - cCARE Fresno, Fresno, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - James Berenson, MD, Inc, West Hollywood, California
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Oncology Specialists, SC, Niles, Illinois
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Vista Oncology, Olympia, Washington